CLINICAL TRIAL: NCT04064203
Title: The Effect of Insulin-induced Hypoglycaemia on Gut-derived Glucagon Secretion
Brief Title: The Effect of Insulin-induced Hypoglycaemia on Gut-derived Glucagon Secretion (Px-Hypo)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Consultant endocrinologist, Professor of, University Hospital, Gentofte, Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-17014216
Record Dates: First submitted 2019-08-16; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Diabetes After Total Pancreatectomy
Keywords: glucagon
MeSH Terms: interventions — Glucose Tolerance Test

STUDY DESIGN:
Intervention Model Description: 12 totally pancreatectomized patients and 12 healthy control subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Totally pancreatectomized patients (Experimental): Oral glucose tolerance test + insulin-induced hypoglycaemic clamp followed by an oral glucose tolerance test
  Interventions: Other: Oral glucose tolerance test; Other: Clamp experiment
- Healthy controls (Experimental): Oral glucose tolerance test + insulin-induced hypoglycaemic clamp followed by an oral glucose tolerance test
  Interventions: Other: Oral glucose tolerance test; Other: Clamp experiment

INTERVENTIONS:
Other: Oral glucose tolerance test — 50 grams OGTT
Other: Clamp experiment — insulin-induced hypoglycaemic clamp followed by an 50 grams OGTT

SUMMARY:
The overall objective of this study is to investigate whether hypoglycaemia (the most potent stimulus of pancreatic glucagon secretion) affects the secretion of gut-derived glucagon in totally pancreatectomized patients.

DETAILED DESCRIPTION:
The investigators want to assess the plasma glucagon response to insulin-induced hypoglycaemia in totally pancreatectomised patients and at the same time evaluate whether hypoglycaemia affects a range of other products from endocrine cells in the gastrointestinal tract including ghrelin, gastrin, cholecystokinin (CCK), glucose-dependent insulinotropic polypeptide (GIP), GLP-1, glucagon-like peptide-2 (GLP-2), oxyntomodulin and peptide YY (PYY). Furthermore the investigators will evaluate how hypoglycaemia in these patients affects other counter-regulatory mechanisms including plasma responses of the hormones adrenaline, noradrenaline, growth hormone and cortisol as well as the rate of gastric emptying rate (which under normal circumstances accelerates during hypoglycaemia) during an oral glucose tolerance test (OGTT).

ELIGIBILITY:
Inclusion Criteria:

Pancreatectomised patients

* Caucasian above 30 years of age who have undergone total pancreatectomy
* Blood haemoglobin >7.0 mmol/l for males and >6.5 mmol/l for females Non-diabetic control subjects
* Normal fasting plasma glucose and normal HbA1c (according to the World Health Organization (WHO) criteria)
* Normal blood haemoglobin
* Caucasian above 30 years of age
* BMI (body mass index) 17-30
* Informed consent

Exclusion Criteria:

Pancreatectomised patients

* Pancreatectomy within the last 3 months
* Ongoing chemotherapy or chemotherapy within the last 3 months
* Previous or ongoing treatment with GLP-1 receptor agonists or dipeptidyl peptidase 4 (DPP-4) inhibitors
* Inflammatory bowel disease
* Gastrointestinal resection (other than the gastro-duodenectomy performed in connection with total pancreatectomy) and/or ostomy
* Nephropathy (eGFR<60 and/or albuminuria)
* Known liver disease (excluding non-alcoholic fatty liver disease) and/or serum alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >3 × normal values)
* Severe lung disease
* Pregnancy and/or breastfeeding
* Age above 85 years
* Uncontrolled hypertension and/or significant cardiovascular disease
* Any condition that the investigator feels would interfere with trial participation Non-diabetic control subjects
* Diabetes or prediabetes (according to WHO criteria)
* First-degree relatives with diabetes
* Inflammatory bowel disease
* Gastrointestinal resection and/or ostomy
* Nephropathy (serum creatinine >150 µmol/l and/or albuminuria)
* Known liver disease (excluding non-alcoholic fatty liver disease) and/or serum ALAT and/or serum ASAT >3 × normal values)
* Severe lung disease
* Pregnancy and/or breastfeeding
* Age above 85 years
* Uncontrolled hypertension and/or significant cardiovascular disease
* Any condition that the investigator feels would interfere with trial participation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
p-glucagon | -30, -15, 0, 15, 40, 50, 60, 70, 80, 90, 105, 120, 135, 150, 165, 180, 210, 240 minutes
  Plasma glucagon excursions measured as incremental area under the curve (iAUC)

SECONDARY OUTCOMES:
p-glucose | -30, -15, 0, 15, 40, 50, 60, 70, 80, 90, 105, 120, 135, 150, 165, 180, 210, 240 minutes
  plasma glucose excursions measured as incremental area under the curve (iAUC)
GIP, GLP-1, GLP-2, GIP, oxyntomodulin, ghrelin, peptide YY, gastrin | -30, -15, 0, 15, 40, 50, 60, 70, 80, 90, 105, 120, 135, 150, 165, 180, 210, 240 minutes
  excursions in Gut hormones measured as incremental area under the curve (iAUC)
catecholamines | -30, -15, 0, 15, 40, 50, 60, 70, 80, 90 minutes
  p-adrenaline and p-noradrenaline, excursions measured as incremental area under the curve (iAUC)
cortisol | -30, -15, 0, 15, 40, 50, 60, 70, 80, 90 minutes
  p-cortisol excursions measured as incremental area under the curve (iAUC)
growth hormone | -30, -15, 0, 15, 40, 50, 60, 70, 80, 90 minutes
  p-growth hormone excursions measured as incremental area under the curve (iAUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Hellerup, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided